CLINICAL TRIAL: NCT05377580
Title: A Multicenter, Randomized, Double-blind, Parallel, Placebo-controlled Phase II Clinical Study to Evaluate the Efficacy and Safety of IBI112 in Patients With Moderate to Severe Active Ulcerative Colitis
Brief Title: A Study to Evaluate IBI112 in the Treatment of Moderate to Severe Active Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIBI112B201
Record Dates: First submitted 2022-05-06; First posted 2022-05-17 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Ulcerative Colitis (UC)
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Period 2 IBI112 dose 4 (Experimental)
  Interventions: Drug: Period 2 IBI112 dose 4
- Period 1 IBI112 Placebo (Placebo Comparator)
  Interventions: Drug: Period 1 IBI112 Placebo
- Period 2 IBI112 dose 3 (Experimental)
  Interventions: Drug: Period 2 IBI112 dose 3; Drug: Period 2 IBI112 Placebo
- Period 1 IBI112 dose 2 (Experimental)
  Interventions: Drug: Period 1 IBI112 dose 2
- Period 2 IBI112 Placebo (Placebo Comparator)
  Interventions: Drug: Period 2 IBI112 Placebo
- Period 1 IBI112 dose 1 (Experimental)
  Interventions: Drug: Period 1 IBI112 Placebo; Drug: Period 1 IBI112 dose 1

INTERVENTIONS:
Drug: Period 1 IBI112 Placebo — Intravenous Injection
  Other Names: Placebo
  Arms: Period 1 IBI112 Placebo; Period 1 IBI112 dose 1
Drug: Period 2 IBI112 dose 3 — Subcutaneous injections
  Other Names: IBI112 dose 3
  Arms: Period 2 IBI112 dose 3
Drug: Period 1 IBI112 dose 1 — Intravenous Injection
  Other Names: IBI112 dose 1
  Arms: Period 1 IBI112 dose 1
Drug: Period 1 IBI112 dose 2 — Intravenous Injection
  Other Names: IBI112 dose 2
  Arms: Period 1 IBI112 dose 2
Drug: Period 2 IBI112 dose 4 — Intravenous Injection
  Other Names: IBI112 dose 4
  Arms: Period 2 IBI112 dose 4
Drug: Period 2 IBI112 Placebo — Subcutaneous injections
  Other Names: Placebo
  Arms: Period 2 IBI112 Placebo; Period 2 IBI112 dose 3

SUMMARY:
To evaluate the efficacy of IBI112 induction therapy in patients with moderate and severe active Ulcerative Colitis (UC) to achieve clinical remission.

DETAILED DESCRIPTION:
This is a phase 2 randomized,double-blind, placebo-controlled study to evaluate the efficacy and safety of IBI112 induction and maintenance therapy in subjects with moderate to severe active ulcerative colitis

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of ulcerative colitis at least 3 months ago, including endoscopy evidence supporting UC and histopathological evidence supporting UC diagnosis;
2. Patients with moderate to severe ulcerative colitis, defined as modified Mayo Score ≥4 and endoscopic score ≥2;
3. Subject must have received at least one prior treatment or first use of a biological agent:

Exclusion Criteria:

1. Diagnosis of ischemic colitis, infectious colitis, radiation colitis, microscopic colitis, uncertain colitis, etc., or crohn's disease;
2. UC lesions were limited to rectum or involved colon < 15cm;
3. Evidence of toxic hirschsprung's disease was found during screening;
4. History or evidence of atypical hyperplasia of the colon, adenomatous polyps (not removed before entering the study) or gastrointestinal tumors;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-06-21 (Actual); Study Completion 2025-08-07 (Actual)

PRIMARY OUTCOMES:
Evaluate the effectiveness of IBI112 in inducing clinical remission in patients with moderately to severely active ulcerative colitis (UC) | week 12
  Percentage of subjects who achieved clinical remission at week 12.

SECONDARY OUTCOMES:
The proportion of participants achieving a clinical response at Week 12. | week 12
  Clinical response is defined as a relative decrease from baseline in the modified Mayo score of ≥30% and ≥2 points, along with a relative decrease in the rectal bleeding subscore of ≥1 point or an absolute subscore of 0 or 1.
The proportion of participants achieving symptomatic relief at Week 12. | week 12
  Symptomatic relief is defined as a stool frequency subscore of 0 or 1 and a rectal bleeding subscore of 0.
The proportion of participants achieving endoscopic remission at Week 12. | week 12
  Endoscopic remission is defined as an endoscopic subscore of 0 or 1 within the modified Mayo score.
The proportion of participants achieving mucosal healing at Week 12. | week 12
  Mucosal healing is defined as endoscopic remission, which means an endoscopic subscore of 0 or 1 within the modified Mayo score, and central Geboes histopathological index remission.
The proportion of participants achieving clinical remission at Week 52 during the maintenance treatment period. | week 52
The proportion of participants achieving clinical response at Week 52 during the maintenance treatment period. | week 52
The proportion of participants achieving symptomatic relief at Week 52 during the maintenance treatment period. | week 52
The proportion of participants achieving mucosal healing at Week 52 during the maintenance treatment period. | week 52
The proportion of participants achieving endoscopic remission at Week 52 during the maintenance treatment period. | week 52
The change from baseline in the Inflammatory Bowel Disease Questionnaire (IBDQ) scores at Week 12, Week 52 during the maintenance treatment period, and Weeks 24 and 64 during the extension treatment period. | Week 12, Week 52，Weeks 24 and 64
The change from baseline in the 36-item Short Form Health Survey (SF-36) scores at Week 12, Week 52 during the maintenance treatment period, and Weeks 24 and 64 during the extension treatment period. | Week 12, Week 52，Weeks 24 and 64

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No